CLINICAL TRIAL: NCT01952691
Title: Initial Effects of Kinesiotaping in Conservative Treatment of Hallux Valgus
Brief Title: Initial Effects of Kinesiotaping in Non Surgical Treatment of Hallux Valgus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, GulOznur KARABICAK, Ms PT, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEK 10/58-48
Record Dates: First submitted 2013-09-19; First posted 2013-09-30 (Estimated); Results first posted 2015-04-06 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2015-04

CONDITIONS: Hallux Valgus; Pain
Keywords: hallux valgus; pain; conservative; treatment
MeSH Terms: conditions — Hallux Valgus; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- kinesiotaping (Experimental): all patients were implemented a kinesiotaping to align the hallux to correct position
  Interventions: Device: kinesiotaping

INTERVENTIONS:
Device: kinesiotaping — correction method was used to align hallux.

SUMMARY:
The main aim of this study was to find the initial effects of kinesiotaping on pain and joint alignment used in the conservative treatment of hallux valgus.

22 female patients diagnosed with hallux valgus participated in this study. Kinesiotaping was implemented after the first assessment and renewed in the 3rd, 7th and 10th days. The main outcome measures were the pain hallux adduction angle. Kinesiotaping may be an effective treatment option in decreasing pain and deformity in hallux valgus deformity who are conservatively treated. In future studies this method might be shown in larger sample groups at longer periods of treatment comparing with alternative treatment approaches like exercise or orthotics.

DETAILED DESCRIPTION:
Hallux valgus is a common pathologic entity affecting the great toe. Taping is an alternative method used to treat hallux valgus. The main aim of this study was to find the initial effects of kinesiotaping on pain and joint alignment used in the conservative treatment of hallux valgus.

22 female patients diagnosed with 13 bilateral, 7 right, 2 left totally 35 with hallux valgus participated in this study. Kinesiotaping was implemented after the first assessment and renewed in the 3rd, 7th and 10th days. The main outcome measures were the change in pain was assessed by using Visual Analogue Scale (VAS) and hallux adduction angle was measured by the universal goniometry. Secondary outcome measures were Patients' functional status was measured by Foot Function Index (FFI) and AOFAS. The plain radiographic results were also measured before and after 1-month of treatment.

Pain and disability was controlled by KinesioTape® implementation in patients with hallux valgus. Kinesiotaping may be an effective treatment option in decreasing pain and deformity in hallux valgus deformity who are conservatively treated. In future studies this method might be shown in larger sample groups at longer periods of treatment comparing with alternative treatment approaches like exercise or orthotics.

ELIGIBILITY:
Inclusion Criteria:

* Hallux adduction angle between 15-40º
* Pain intensity higher than 5 according to VAS
* 20- 45 years age female
* No trauma, surgery history
* Surgery is indicated but the patient is willing to try conservative treatment options

Exclusion Criteria:

* Fracture, surgery history on the great toe
* Systematic disease (Rheumatoid Arthritis, Systematic Lupus Erythematosus Diabetes)
* Using NSAID, analgesic drug
* Hallux rigidus diagnosis

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2011-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: nilgun bek, Phd PT, Study Director — Hacettepe University; Ugur TIFTIKCI, MD, Study Chair — beypazari hospital; Gul Oznur KARABICAK, MS PT, Principal Investigator — Hacettepe University

RESULTS

PARTICIPANT FLOW:
Groups:
- Kinesiotaping Implementation: kinesiotaping was implemetedto all patients to align the hallux to correct position for 10 days. Each patient was re-assessed and the taping implementation was renewed on the 3rd, 7th and 10th days of the treatment.
  kinesiotaping: correction method was used to align hallux's adduction position.
Period: Overall Study
Arm/Group | Kinesiotaping Implementation
Started | 22
Completed | 20
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Kinesiotaping
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Adduction Angle of Hallux With X RAY
Description: X ray was obtained in non-weight bearing sitting position. It's aimed to see the treatment effects kinesio taping
Time Frame: up to 30 days after the treatment
Population: 35 feet's X Ray results were obtained from 22 patients before treatment protocol was performed.
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: feet
Arm/Group | Kinesiotaping Implementation
Number analyzed (Participants) | 22
Number analyzed (feet) | 35
degrees
  before treatment protocol | 22.6 (5.0)
  after treatment was ceased | 19.3 (5.3)

2. Secondary Outcome: FFI
Description: We aimed to see the change in functional status with FFI (Foot function index) scale The FFI is a self-administered index consisting of 23 items divided into 3 sub-scales used to score each question on a scale from 0 (no pain or difficulty) to 10 (worst pain imaginable or so difficult it required help) that best describes the patients' foot over the past week. Patients were instructed to mark a VAS score for each question. The total score was calculated using only the questions answered.
Time Frame: baseline, on the 3rd, 7th, 10th and 30th days during the treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: feet
Arm/Group | Kinesiotaping Implementation
Number analyzed (Participants) | 22
Number analyzed (feet) | 35
units on a scale
  before treatment protocol | 3.2 (1.6)
  after treatment was ceased (30th day) | 0.84 (1.24)

3. Secondary Outcome: Adduction Angle
Description: we aimed to see the change in hallux valgus angle during treatment.
Time Frame: baseline and 30th days.
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: feet
Arm/Group | Kinesiotaping Implementation
Number analyzed (Participants) | 22
Number analyzed (feet) | 35
degrees
  before treatment protocol | 20.2 (4.7)
  after treatment was ceased (30th day) | 14.3 (5.0)

ADVERSE EVENTS:
Arm/Group | Kinesiotaping Implementation
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes